CLINICAL TRIAL: NCT02263833
Title: Post Marketing Surveillance of Mircera®
Brief Title: An Observational, Prospective, Safety Study of Mircera (Monopegylated Epoetin Beta) in Clinical Practice
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML22560
Record Dates: First submitted 2014-10-08; First posted 2014-10-13 (Estimated); Results first posted 2016-07-28 (Estimated); Last update posted 2016-09-07 (Estimated); Status verified 2016-07

CONDITIONS: Kidney Disease, Chronic
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Overall Participants: Participants not previously on erythropoietin-stimulating agent (ESA) therapy and participants on ESA therapy who were switched to Mircera
  Interventions: Drug: Mircera

INTERVENTIONS:
Drug: Mircera — Participants received Mircera according to individualized physician-prescribed regimen.

SUMMARY:
This national study was a post-marketing surveillance study conducted in Korea from 29 August 2008 to 28 August 2012 to meet local regulatory requirements for Mircera (monopegylated-epoetin beta). Prospective participant-based data collection was evaluated for safety/risk assessments and effectiveness. No specific study-related procedures are required. Participants were to be followed up as long as possible at the physician's discretion.

ELIGIBILITY:
Inclusion Criteria:

* Adult, aged >18 years
* Participants with stage 3-5 chronic kidney disease and hemodialyzed participants
* Signed informed consent

Exclusion Criteria:

* Current participation in a clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with chronic renal anemia regardless of pre-dialysis / dialysis in Korea. Participants who were prescribed Mircera by their physician according to the local Korean Mircera label, for the treatment of anemia associated with chronic kidney disease who require ESA therapy could be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 748 (Actual)
Dates: Start 2009-09; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In total, 748 participants were enrolled from 27 sites, of which only 742 participants were used for safety and efficacy analysis.
Groups:
- Overall Participants: Participants not previously on erythropoietin-stimulating agent (ESA) therapy and participants on ESA therapy who were prescribed Mircera either subcutaneously (SC) or intravenously (IV) according to local Korean Mircera label and at physician's discretion were observed as per physician's discretion, approximately up to 4 years.
Period: Overall Study
Arm/Group | Overall Participants
Started | 742
Completed | 742
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Participants: Participants not previously on ESA therapy and participants on ESA therapy who were prescribed Mircera either SC or IV according to local Korean Mircera label and at physician's discretion were observed as per physician's discretion, approximately up to 4 years.
Arm/Group | Overall Participants
Number analyzed (Participants) | 742
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 376
  Male | 366

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Adverse Event (AE) and a Serious Adverse Event
Description: An AE was defined as any untoward medical occurrence in a participant administered with Mircera and which does not necessarily have a causal relationship with Mircera. A Serious Adverse Event (SAE) is any experience that suggests a significant hazard, contraindication, side effect or precaution. It is any AE that at any dose fulfills at least one of the following criteria: is fatal; is life threatening; requires in-patient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; is medically significant or requires intervention to prevent one or other of the outcomes listed above.
Time Frame: At physician's discretion, up to 4 years
Population: Safety population included all participants who received at least a dose of Mircera and had the safety assessment at least once.
Measure: Number; unit: percentage of participants
Arm/Group | Overall Participants
Number analyzed (Participants) | 742
percentage of participants
  Adverse event | 3
  Serious adverse event | 0.40

2. Primary Outcome: Percentage of Participants With an Adverse Drug Reaction (ADR)
Description: ADRs were defined as any response to a drug which was noxious and unintended, and which occurred at dose normally used related to the pharmacological properties. It was defined as any AE categorized as "definitely related","probably related", "possibly related", and "unknown" by investigators. In case that an ADR was not written on local Korean Mircera label, it was classified as "Unexpected". An AE was defined as any untoward medical occurrence in a participant administered with Mircera and which does not necessarily have a causal relationship with Mircera.
Time Frame: At physician's discretion, up to 4 years
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Overall Participants
Number analyzed (Participants) | 742
percentage of participants | 2.0

3. Other Pre Specified Outcome: Percentage of ESA Naïve Participants Having an Increase in Hemoglobin (Hb) Level of at Least 1 g/dL From Baseline and Reaching the Hb Level Greater Than or Equal to (>/=) 11 g/dL Without Red Blood Cell Transfusion
Time Frame: Up to 4 years
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Percentage of Participants on ESA Therapy Who Were Switched to Mircera Having a Hemoglobin Concentration in the Range of 10 to 12 g/dL
Time Frame: Up to 4 years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 4 years
Description: An AE was defined as any untoward medical occurrence in a participant administered with Mircera and which does not necessarily have a causal relationship with Mircera.
Arm/Group | Overall Participants
Serious Adverse Events (participants affected / at risk) | 3/742
Other Adverse Events (participants affected / at risk) | 0/742
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Participants (N=742)
Atrioventricular block (Cardiac disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.